CLINICAL TRIAL: NCT01884948
Title: A Randomized, Double-blind Study of the Effects of Omega-3 Fatty Acids (Omegaven™) on Outcome After Major Liver Resection
Brief Title: Effects of Omega-3 Fatty Acids on Outcome After Major Liver Resection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: Omegaven - Zurich
Record Dates: First submitted 2013-06-14; First posted 2013-06-24 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Major Liver Surgery
Keywords: at least 1 segment; multiple wedge resections (≥3)
MeSH Terms: interventions — fish oil triglycerides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omegaven™ (Active Comparator): Omegaven™ (approval number:54750 Swissmedic)- 100ml intravenously. The first dose (Omegaven™ or placebo) is administered in the evening before surgery, the second dose at the beginning of anesthesia. The maximum infusion rate must be adjusted to bodyweight (0.5 ml Omegaven™/kg/hour).
  Interventions: Drug: Omegaven™
- NaCl 0.9% (Placebo Comparator): 100ml of saline is used as a placebo comparator and administered as described above.

INTERVENTIONS:
Drug: Omegaven™
  Arms: Omegaven™

SUMMARY:
To study the efficacy and safety of intravenous Omegaven™ (vs. Placebo) in reducing postoperative morbidity and mortality after major liver resection.

DETAILED DESCRIPTION:
With two single doses of Omegaven (pre- and postoperatively) we aim to reduce postoperative complications measured by the CCI (Comprehensive Complication Index) and the Clavien Dindo classification of surgical complications. The study will include adults (more than 18 years) patients requiring liver resection of at least 1 segment or multiple wedge resections (≥3).

ELIGIBILITY:
Inclusion criteria:

* Requiring liver resection of at least 1 segment or multiple wedge resections (=3)
* > 18 years of age
* No coagulopathy (INR < 1.2, platelets >150'000 x10E3/µl)
* Understands local language

Exclusion criteria:

* Liver resections <1 segment
* Wedge resections (<3)
* Liver cirrhosis
* Coagulopathy (INR > 1.2, platelets < 150'000 x10E3/µl)
* Hypertriglyceridemia (> 5.0 mmol/l)
* Hypersensitivity or allergy to Omegaven™ or any fish oil or lipid emulsions
* Known allergy to egg protein
* Pregnancy
* Nursing women
* Renal failure(estimated GFR < 30 ml/min/1.73m2)
* Medication impairing platelets aggregation
* Cannot understand local language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | 1 month after hospital discharge
  Complications will be assessed using the Comprehensive Complication Index (CCI) and the Clavien-Dindo complication classification.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Alain Clavien, MD PhD, Principal Investigator — University Hospital Zurich, Visceral and Transplantation Surgery
Locations (1):
- University Hospital Zurich, Visceral and Transplantation Surgery, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Linecker M, Botea F, Aristotele Raptis D, Nicolaescu D, Limani P, Alikhanov R, Kim P, Wirsching A, Kron P, Schneider MA, Tschuor C, Kambakamba P, Oberkofler C, De Oliveira ML, Bonvini J, Efanov M, Graf R, Petrowsky H, Khatkov I, Clavien PA, Popescu I. Perioperative omega-3 fatty acids fail to confer protection in liver surgery: Results of a multicentric, double-blind, randomized controlled trial. J Hepatol. 2020 Mar;72(3):498-505. doi: 10.1016/j.jhep.2019.10.004. Epub 2019 Oct 15. PMID 31626819
- [Derived] Linecker M, Limani P, Botea F, Popescu I, Alikhanov R, Efanov M, Kim P, Khatkov I, Raptis DA, Tschuor C, Beck-Schimmer B, Bonvini J, Wirsching A, Kron P, Slankamenac K, Humar B, Graf R, Petrowsky H, Clavien PA. "A randomized, double-blind study of the effects of omega-3 fatty acids (Omegaven) on outcome after major liver resection". BMC Gastroenterol. 2015 Aug 14;15:102. doi: 10.1186/s12876-015-0331-1. PMID 26268565
- See also: Omegaven — http://www.kompendium.ch/mpro/mnr/8980/html/de